CLINICAL TRIAL: NCT04706910
Title: 18F-DOPA II - PET Imaging Optimization
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00100294
Record Dates: First submitted 2020-12-21; First posted 2021-01-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Congenital Hyperinsulinism; Neuroblastoma; Parkinson Disease; Lewy Body Disease; Neuroendocrine Tumors; Brain Tumor
MeSH Terms: conditions — Congenital Hyperinsulinism; Neuroblastoma; Parkinson Disease; Lewy Body Disease; Neuroendocrine Tumors; Brain Neoplasms | interventions — fluorodopa F 18; Furosemide; 4-chloro-N-(2-furylmethyl)-5-sulfamoylanthranilic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DOPA injection (Experimental): All enrolled participants will receive an intravenous injection of the investigational 18F-DOPA radiopharmaceutical
  Interventions: Drug: 18F-DOPA; Drug: Furosemide Injection

INTERVENTIONS:
Drug: 18F-DOPA — All participants will receive an intravenous injection of 18F-DOPA (4MBq/kg; minimum 110 MBq, maximum 600 MBq) for this study
  Other Names: 18F-dihydroxyphenylalanine
Drug: Furosemide Injection — Some participants will receive an intravenous injection of furosemide (40mg, single dose)
  Other Names: 4-chloro-N-furfuryl-5-sulfamoylanthranilic acid

SUMMARY:
A single centre non-randomized, non-blinded phase III prospective cohort study of 18F-DOPA PET/CT imaging in specific patient populations:

1. Pediatric patients (less than 18 years old) with congenital hyperinsulinism.
2. Pediatric patients (less than 18 years old) with neuroblastoma.
3. Pediatric (less than 18 years old) or Adult patients (18 or older) with known or clinically suspected neuroendocrine tumor.
4. Adult patients (18 or older) with a clinical suspicion of Parkinson's disease or Lewy body dementia.
5. Pediatric (less than 18 years old) or Adult patients (18 or older) with brain tumors.

Image optimization (the primary study objective) and gallbladder activity pattern (the secondary objective) will be evaluated.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

6-[18F]fluoro-dihydroxyphenylalanine (18F-DOPA) is a large neutral amino acid that resembles natural L-3.4-dihydroxyphenylalanine (L-DOPA) biochemically. L-DOPA is a precursor for dopamine, epinephrine (adrenaline), and norepinephrine (noradrenaline), collectively known as catecholamines. 18F-DOPA enters the biochemical pathway of L-DOPA both in the brain and peripherally, and can be imaged with a positron emission tomography / computed tomography (PET/CT) scanner. 18F-DOPA can therefore allow imaging of the L-DOPA metabolic pathway with a high target-to-background ratio providing valuable information for a number of diseases.

While 18F-DOPA is an established diagnostic tracer at a number of different institutions globally, given the short half-life of 18F (110 minutes) this tracer cannot be imported for local use. The Edmonton PET Centre has recently developed a production method for this tracer allowing local access. An initial study at the University of Alberta (Pro00055342) has demonstrated this tracer to have an acceptable safety profile, an expected biodistribution (both physiologic and disease-related), and has established clinical efficacy of the tracer.

In March, 2020 the University of Alberta Hospital (UAH) installed a new PET/CT scanner (GE Discovery MI) with a digital detector system and new iterative image reconstruction algorithms that represent a substantial technological improvement compared to the previously installed scanner. It is expected that this new system will reduce artifact and will increase the sensitivity for the detection of smaller lesions.

Our initial study demonstrated rapid urinary excretion with intense collection of activity within the urinary bladder. While this physiology was expected, it did result in diminished image quality in the evaluation of the pelvis in some patients. Improved image reconstruction algorithms available on the new GE Discovery MI PET/CT system may improve imaged quality related to this problem. Based on our experience with 18F-fluorodeoxyglucose (FDG) PET/CT scans, the administration of intravenous furosemide prior to imaging can also substantially improve the image quality in the pelvis. These potential improvements have not yet been established with 18F-DOPA.

A second observation from our initial study was that many participants demonstrated intense early activity at the gallbladder fundus. While biliary and gallbladder activity are described in the normal biodistribution of 18F-DOPA, the observed distribution suggests that the gallbladder fundus activity reflects primary uptake rather than reflux of activity within bile into the gallbladder.

The rationale for this study is to explore the efficacy of these optimization parameters (new digital PET/CT camera system and use of intravenous furosemide) in the context of 18F-DOPA PET/CT imaging for patients with clinical indications for the scan. Imaging data from this study will be compared with data from the prior study (Pro00055342) to determine if the new digital detector PET/CT technology and preparatory furosemide administration improves image quality for these patients.

A subgroup will also be scanned dynamically at the abdomen to better assess the pattern of gallbladder activity over time. This will include a mixture of clinical indications listed within the inclusion criteria. All patients will be screened for a history of previous gallbladder disease at the time of the scan by questionnaire. The intention of this sub-study is to better determine 18F-DOPA activity patterns associated with the gallbladder and to explore if there is a correlation between dopaminergic degeneration in the brain and the gallbladder.

PURPOSE AND STUDY OBJECTIVE:

Trial Type: Phase III non-randomized, non-blinded prospective cohort clinical trial of patients with a clinical indication for 18F-DOPA PET/CT imaging.

The primary purpose of this study is to assess optimization parameters for 18F-DOPA PET CT imaging at UAH including the impact of new digital detector PET/CT technology as well as the impact of preparatory intravenous furosemide administration on image quality within the pelvis. A secondary purpose of this study is to better delineate the pattern of 18F-DOPA activity associated with the gallbladder and to explore if there is a relationship between dopaminergic denervation in the gallbladder and the brain.

Only patient populations for which there are established clinical indications for the use of 18F-DOPA will be included in this study. Participation in this study will allow access to this tracer for patients in Alberta as there is no Health Canada approved similar tracer currently available. 18F-DOPA is an established clinical tracer at multiple institutions globally and has been approved for clinical use at multiple European centres for many (10+) years. Established clinical indications in the literature include:

1. Pediatric patients (less than 18 years old) with congenital hyperinsulinism. The 18F-DOPA scan is used to plan required surgical intervention for these patients.
2. Pediatric patients (less than 18 years old) with neuroblastoma. The 18F-DOPA scan is indicated for pre-operative assessment of a mass suspected to be a neuroblastoma, staging, re-staging, and assessment of recurrence in this patient group.
3. Pediatric (less than 18 years old) or Adult patients (18 or older) with known or clinically suspected neuroendocrine tumor. These include patients with carcinoid tumor, pheochromocytoma, paraganglioma, and medullary thyroid cancer. 18F-DOPA is indicated for metabolic assessment of a mass suspected to represent one of these tumor-types, for staging of a known tumor, for re-staging, and for assessment of recurrence in this patient group.
4. Adult patients (18 or older) with a clinical suspicion of Parkinson's disease or Lewy body dementia. 18F-DOPA is indicated to differentiate benign essential tremor from Parkinson's disease in this patient group [22-26]. 18F-DOPA may also be used to differentiate Lewy body dementia from other dementia types.
5. Pediatric (less than 18 years old) or Adult patients (18 or older) with brain tumors (primary or metastatic). 18F-DOPA is indicated for biopsy planning, radiation therapy planning, and post-therapy assessment to differentiate residual viable tumor from post-therapy necrosis in this patient population.

When requested for patients falling into one of these diagnostic groups, an 18F-DOPA PET/CT scan will be performed and interpreted clinically with the results conveyed to the referring physician.

Image optimization (the primary study objective) will be evaluated based on the following:

* For patients with abnormal activity, the smallest 3 lesions will be recorded in terms of size (mm) and activity (SUVmax). For PET-avid lesions, the size measurement will be based on measuring the maximum dimension of the corresponding lesion on the CT scan component if possible. If not possible, a size measurement based on the PET images will be used. The minimum lesion size and average (3 smallest lesions) will be compared with a cohort of scans acquired on the previous non-digital PET/CT scanner (retrospective cohort of 50 positive patients, Pro00055342).
* The SUVmax, SUVmean, and SUV standard deviation of urinary bladder activity will be measured and compared to a retrospective cohort of 50 patients from a previous study (Pro00055342)
* A subjective score will be applied to the pelvis with respect to image artifact related to bladder activity (0 = no artifact, 1 = mild artifact, 2 = severe artifact). This will be compared to scoring of the previous study (retrospective cohort of 50 patients, Pro00055342) retrospectively.

Gallbladder activity pattern (the secondary objective) will be evaluated based on the following:

* SUVmax measurements of the gallbladder fundus, gallbladder neck, common bile duct, right and left main intrahepatic ducts, and liver parenchyma (right and left lobes, 3 cm diameter VOI) will be measured at 5 minute increments. These will be analyzed in total, and subgroups will be compared (32 PD vs. 32 non-PD participants).
* All participants will be screened by questionnaire at the time of the scan as to whether there is a history of previous gallbladder disease. The positive response rate will be compared between three groups: non-PD patients, PD patients with objective evidence of dopaminergic denervation (positive FDOPA scan), PD patients without objective evidence of dopaminergic denervation (negative FDOPA scan).

PATIENT POPULATION:

A total of 800 patients who meet the inclusion criteria will be identified based on referrals from physicians who deem the imaging studies potentially useful for clinical care. It is anticipated that complete enrollment will take 5 years (approximately 160 scans per year).

Sample size calculation is based on the following. There will typically be 5 participants total scanned per day. Dynamic imaging will be restricted to one patient per scanning day due to time constraints related to the scanner, as this requires the participant to lie quietly in the PET/CT scanner for up to one hour. Allowing for this restriction, it is estimated that the overall participation rate for dynamic scanning will be 10%. Based on a minimum total sample size of 64 participants for the secondary objective analysis, a total minimum study population of 640 is required. Allowing for some potential buffer for recruitment, a total of 800 participants is planned.

The minimum sample size of 64 participants is based on the following estimations: gallbladder fundus SUVmax mean 10.9, SUVmax DS 4.6 (measured from cohort of 10 patients from the previous study), α = 0.05, and power = 0.80. Two groups of 32 participants (64 total) should allow for detection of a minimum 30% difference in SUVmax involving the gallbladder fundus between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients (less than 18 years old) with congenital hyperinsulinism.
2. Pediatric patients (less than 18 years old) with neuroblastoma.
3. Pediatric (less than 18 years old) or Adult patients (18 or older) with known or clinically suspected neuroendocrine tumor.
4. Adult patients (18 or older) with a clinical suspicion of Parkinson's disease or Lewy body dementia.
5. Pediatric (less than 18 years old) or Adult patients (18 or older) with brain tumors.

Exclusion Criteria:

1. Unable to obtain consent
2. Weight >225 kg (weight limitation of PET/CT scanner)
3. Adult patients unable to lie flat for 20-30 minutes to complete the PET-CT session.
4. Young pediatric patients (less than 13 years old) who are unable to lie flat for 20-30 minutes and for whom clinical sedation is contraindicated (as determined by a pediatric anaesthesiologist).
5. Lack of intravenous access
6. History of previous cholecystectomy (excluded from dynamic abdomen sub-study only)
7. Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Minimum lesion detectibility (size) | Within 1 month of PET/CT scan
  Measurement of size (mm) of the three smallest lesions
Assessment of bladder activity | Within 1 month of PET/CT scan
  Measurement of standardized uptake value (SUV) for urinary bladder activity
Assessment of bladder activity artifact | Within 1 month of PET/CT scan
  Subjective scoring (0-2 scale) of image artifact in pelvis related to bladder activity
Minimum lesion detectability (SUV) | Within 1 month of PET/CT scan
  Measurement of the standardized uptake value (SUV) of the three smallest lesions

SECONDARY OUTCOMES:
Gallbladder activity pattern | Within 3 months of PET/CT scan
  Assessment of SUVmax of various segments of the biliary tree at different time points after 18F-DOPA injection using a subgroup of participants (64 total)
Gallbladder disease questionnaire | At the time of enrollment
  All participants will complete a questionnaire regarding a history of gallbladder disease

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Abele, MD, Principal Investigator — University of Alberta
Locations (1):
- WC Mackenzie Health Science Centre / University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No